CLINICAL TRIAL: NCT07281638
Title: Bedside Bike Early Mobilization Program for Inpatients
Acronym: BB-STEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Babar Khan, MD, MS, Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 28224
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Immobility Syndrome; Deep Venous Thrombosis; Delirium; Hospital Acquired Condition; Fall; Mobility Limitation
Keywords: Immobility Harm; Hospital-Acquired Disability; Falls; Deconditioning; In-bed exercise
MeSH Terms: conditions — Venous Thrombosis; Delirium; Iatrogenic Disease; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention Group (receiving Bedside Bike + Usual Care) (Experimental): All enrolled participants receive the Bedside Bike device plus standard hospital care. Installed within 24 hours of admission, patients are trained on device operation and safety. Setup takes <1 minute. Patients use the device daily throughout hospitalization, targeting ≥15 minutes per session. Exercise is self-paced with adjustable resistance via patient-controlled dial. Recumbent (in-bed) cycling allows unsupervised, patient-initiated use without staff presence. Average duration is 5-7 days (enrollment to discharge). Participants continue all standard care including physical/occupational therapy, ambulation, medications, and nutrition.
  Interventions: Device: Bedside Bike

INTERVENTIONS:
Device: Bedside Bike — The Bedside Bike is a Class I medical device (21 CFR §890.5370, product code ION) featuring a magnetic resistance mechanism powering arm and leg pedal systems with a universal clamp for standard hospital bed frames. Key safety features include smooth surfaces without sharp edges, immediate stop mechanism with no momentum carry-over, cushioned pedals supporting single-pedal operation for hemiparesis, self-retracting tether cable preventing entanglement, battery-powered operation eliminating tripping hazards, nearly silent operation, lightweight construction, and soft-start/soft-stop resistance adjustment.

SUMMARY:
Hospital immobility leads to serious complications including muscle loss, weakness, delirium, pressure ulcers, and blood clots. Despite being medically stable, hospitalized patients spend over 90% of their time in bed due to staffing shortages, fall risks, and limited physical therapy availability. Within one week of admission, patients can lose approximately 2% of thigh muscle mass per day, and nearly half develop clinically significant hospital-acquired weakness.The Bedside Bike is a portable, low-resistance exercise device that clamps securely to hospital beds, allowing patients to perform leg and arm cycling exercises safely without leaving their bed. This study will evaluate whether hospitalized patients at Indiana University Health facilities can feasibly and safely use the Bedside Bike to maintain mobility during their hospital stay.This quality improvement study will enroll 80 adult inpatients expected to stay at least 3 days. All participants will receive the Bedside Bike in addition to usual care (standard physical therapy and medical treatment). The study will measure how often patients use the device, whether it is safe (tracking any device-related problems), and whether it may help improve outcomes such as hospital length of stay, functional mobility scores, discharge to home, and rates of hospital-acquired weakness. Participants will have functional assessments at admission and discharge, use the Bedside Bike throughout their hospitalization (targeting at least 15 minutes daily), and be followed for 60 days after discharge to track readmissions, falls, living arrangements, and mortality.

DETAILED DESCRIPTION:
Background and Rationale:

Immobility during hospitalization is a widespread and often preventable cause of disability, particularly among older adults and patients recovering from critical illness. Research demonstrates that very modest activity confers significant benefits: walking just 275 steps per day reduces 30-day readmissions by 10% in older inpatients, and a single 20-minute cycling session on weekdays shortens length of stay and improves functional recovery in ventilated ICU patients. However, most patients remain largely immobile despite being physiologically capable of low-intensity exercise.

The Bedside Bike addresses key barriers to inpatient mobility by eliminating the need to transfer out of bed (reducing fall risk), requiring less than 1 minute of staff setup time (addressing staffing constraints), providing adjustable resistance for progressive exercise, and allowing patients to exercise independently without navigating hallways with IV lines and catheters. The device is FDA-cleared (Class I, product code ION, 21 CFR §890.5370) and has been tested with healthcare providers and healthy volunteers without safety concerns.

Study Design and Implementation:

This is a prospective, single-arm quality improvement implementation study conducted across three Indiana University Health hospital units: IU Methodist Post-ICU step-down unit, IU Bloomington ortho/neuro and medical/surgical units, and IU North medical/surgical unit. The study uses a pragmatic design embedded within routine clinical care, with contemporaneous historical unit-level metrics from 2025 serving as comparison benchmarks.

Device Setup and Operation:

After informed consent, the Bedside Bike is installed at the bedside and patients receive training on its use. The device clamps securely to the bed frame with pedals positioned approximately 10 cm above the mattress. Patients can adjust resistance via a dial and exercise at their own pace, targeting at least one 15-minute session daily. A quick-release lever allows the device to be disengaged in under 2 seconds if needed for patient transfers or clinical procedures.

The Bedside Bike includes a Bluetooth-enabled telemetry module that automatically records exercise metrics including duration, revolutions per minute, and resistance level. Data is encrypted and uploaded nightly to a secure REDCap database at Indiana University. Between patients, the device is cleaned with standard hospital disinfectant, and Clinical Engineering performs weekly quality assurance checks.

Integration with Standard Care:

Patients continue all standard medical care without restrictions. Physical therapy, occupational therapy, and progressive ambulation programs proceed as usual. The Bedside Bike is designed to augment-not replace-skilled therapy sessions. There are no restrictions on pain medications, sleep aids, or nutritional support. Cycling is temporarily paused during hemodialysis or when telemetry alarms require clinical attention.

Data Safety Monitoring:

The Principal Investigator leads weekly data safety monitoring huddles to review enrollment progress, device utilization patterns, and adverse events. Any unanticipated serious adverse event triggers immediate IRB notification within 48 hours. The study protocol includes automatic pause criteria: enrollment halts if any device-related serious adverse event occurs or if feasibility drops below 40% for two consecutive weeks, pending comprehensive safety review.

Duration and Follow-up:

The enrollment period spans 3 months (February through April 2026) with approximately 16 patients enrolled monthly across all sites. Each participant is followed through hospital discharge plus 60 days post-discharge. The final 60-day follow-up is completed by the end of June 2026, with database lock and analysis extending through September 2026.

Statistical Design:

With N=80 participants, the study provides 90% power (α=0.05, two-tailed, assuming SD of 2 days) to detect a clinically meaningful 0.2-day reduction in length of stay compared to historical unit averages. This sample size accounts for potential dropouts and incomplete data. Missing data under 5% will be handled using multiple imputation (m=5 iterations); higher rates of missingness will default to complete-case analysis.

This pragmatic feasibility study will provide critical data on device utilization, safety profile, and preliminary effectiveness signals to inform the design of larger randomized controlled trials and guide clinical implementation strategies for in-bed cycling technology across diverse inpatient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Admitted to participating hospital unit within 24 hours or less
* Expected hospital stay of at least 3 days
* Able to follow one-step commands
* Anti-gravity leg strength
* Informed consent obtained from patient or legally authorized representative

Exclusion Criteria:

* Hemodynamic instability requiring vasopressor support with systolic blood pressure <90 mmHg
* Requiring fraction of inspired oxygen (FiO₂) >0.6 or positive end-expiratory pressure (PEEP) >8 cm H₂O
* Uncontrolled cardiac arrhythmia
* Open lower extremity wounds within the pedal arc area
* Lower limb fracture requiring traction or immobilization
* Active deep vein thrombosis (DVT) without therapeutic anticoagulation
* Body mass index (BMI) >45 kg/m² (exceeds device reach limit)
* Current pregnancy
* Concurrent enrollment in another interventional clinical trial that would conflict with study procedures or outcomes

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Device Utilization Feasibility | First 5 hospital days (or until discharge if sooner)
  Percentage of enrolled participants who achieve at least 75 cumulative minutes of Bedside Bike use during their first 5 hospital days. Success criterion: ≥80% of participants meet this threshold.
Incidence of Device-Related Adverse Events | From enrollment through hospital discharge, approximately 5-7 days on average
  Rate of device-related adverse events (AEs) and serious adverse events (SAEs). Safety success criteria: zero device-related SAEs and ≤5% rate of minor device-related AEs. Device-related events are defined as any adverse outcome directly attributable to the Bedside Bike device itself or its use.
Hospital Length of Stay | From hospital admission to discharge, approximately 5-7 days on average
  Duration of index hospitalization in days, compared to 2025 unit-specific median length of stay. Target: reduction of ≥0.2 days versus historical benchmark.

SECONDARY OUTCOMES:
Change in AM-PAC 6-Clicks Mobility Score | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in Activity Measure for Post-Acute Care (AM-PAC) "6 Clicks" Basic Mobility Inpatient Short Form score from baseline to discharge. Target: improvement of ≥2 points. Score range 6-24, with higher scores indicating better mobility function.
Change in AM-PAC 6-Clicks Activities of Daily Living Score | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in Activity Measure for Post-Acute Care (AM-PAC) "6 Clicks" Activities of Daily Living (ADL) Inpatient Short Form score from baseline to discharge. Score range 6-24, with higher scores indicating better ADL function.
Discharge Disposition to Home | At hospital discharge, approximately 5-7 days after admission
  Percentage of participants discharged directly home (versus inpatient rehabilitation facility, skilled nursing facility, long-term acute care hospital, or death). Target: increase of ≥7% compared to 2025 unit-specific historical rate.
Incidence of Hospital-Acquired Weakness | At hospital discharge, approximately 5-7 days after admission
  Percentage of participants with hospital-acquired weakness defined as Medical Research Council (MRC) sum score <48 at discharge. MRC sum score assesses strength in 12 muscle groups bilaterally (range 0-60), with scores <48 indicating clinically significant weakness. Target incidence: <30%.
New Institutionalization at 60 Days Post-Discharge | 60 days post-hospital discharge
  Percentage of participants requiring new placement in skilled nursing facility, long-term care facility, or inpatient rehabilitation facility at 60 days post-discharge (among those discharged home initially).
Change in One-Minute Sit-to-Stand Repetitions | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in number of sit-to-stand repetitions completed in one minute from baseline to discharge. This test measures lower extremity strength and functional capacity.
Change in Six-Minute Walk Test Distance | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in distance walked in six minutes from baseline to discharge, measured in meters. This test assesses cardiorespiratory fitness and functional exercise capacity.
Change in EQ-5D Quality of Life Score | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in EQ-5D (EuroQol 5-Dimension) health-related quality of life score from baseline to discharge. The EQ-5D assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in HADS total score from baseline to discharge. HADS consists of anxiety and depression subscales (each 0-21, total 0-42), with higher scores indicating greater symptom severity.
Change in Berg Balance Scale Score | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in Berg Balance Scale score from baseline to discharge. Scale ranges 0-56, with higher scores indicating better balance. Scores <45 indicate higher fall risk.
Change in Timed Up and Go Test Duration | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in time (seconds) required to stand from a chair, walk 3 meters, turn around, walk back, and sit down from baseline to discharge. Shorter times indicate better functional mobility.
Change in Quadriceps Isometric Strength | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in quadriceps muscle strength measured via handheld dynamometry from baseline to discharge, measured in kilograms of force or Newtons.
Change in Johns Hopkins Highest Level of Mobility (JH-HLM) Score | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in JH-HLM score from baseline to discharge. Scale ranges 1-8, with higher scores indicating greater mobility independence (1=lying in bed to 8=ambulating >250 feet).
Change in Estimated VO2 Max | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in estimated maximal oxygen consumption (VO2 max) from baseline to discharge, measured in mL/kg/min. VO2 max indicates cardiorespiratory fitness.
Change in Braden Skin Score | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in Braden Scale for Predicting Pressure Sore Risk from baseline to discharge. Scale ranges 6-23, with lower scores indicating higher risk for pressure ulcer development.
Change in Morse Fall Scale Score | Baseline (within 24 hours of admission) to discharge (approximately 5-7 days)
  Change in Morse Fall Scale score from baseline to discharge. Scale ranges 0-125, with higher scores indicating greater fall risk (0-24=low risk, 25-50=moderate risk, ≥51=high risk).
60-Day Hospital Readmission Rate | 60 days post-hospital discharge
  Percentage of participants readmitted to any hospital within 60 days of discharge from index hospitalization, assessed via medical record review.
Incidence of Falls Within 60 Days Post-Discharge | 60 days post-hospital discharge
  Number and percentage of participants experiencing one or more falls after hospital discharge, occurring in any setting (home, post-acute care facility, or community), assessed via medical record review and telephone follow-up.
60-Day All-Cause Mortality | 60 days post-hospital discharge
  All-cause mortality within 60 days of hospital discharge, assessed via medical record review and telephone follow-up.
Living Setting at 60 Days Post-Discharge | 60 days post-hospital discharge
  Participant's living arrangement at 60 days post-discharge, categorized as: home (independent), home (with assistance), skilled nursing facility, long-term care facility, inpatient rehabilitation, other, or deceased.
Total Healthcare Costs Through 60 Days | From hospital admission through 60 days post-discharge (approximately 65-75 days total)
  Total direct healthcare costs including index hospitalization and all healthcare utilization within 60 days post-discharge, obtained from de-identified aggregated claims data. Costs measured in US dollars.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gales, DPT, Principal Investigator — Indiana University; Babar Khan, MD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Regenbogen SE, Cain-Nielsen AH, Syrjamaki JD, Chen LM, Norton EC. Spending On Postacute Care After Hospitalization In Commercial Insurance And Medicare Around Age Sixty-Five. Health Aff (Millwood). 2019 Sep;38(9):1505-1513. doi: 10.1377/hlthaff.2018.05445. PMID 31479364
- [Background] Brown CJ, Friedkin RJ, Inouye SK. Prevalence and outcomes of low mobility in hospitalized older patients. J Am Geriatr Soc. 2004 Aug;52(8):1263-70. doi: 10.1111/j.1532-5415.2004.52354.x. PMID 15271112
- [Background] Brown CJ, Redden DT, Flood KL, Allman RM. The underrecognized epidemic of low mobility during hospitalization of older adults. J Am Geriatr Soc. 2009 Sep;57(9):1660-5. doi: 10.1111/j.1532-5415.2009.02393.x. Epub 2009 Aug 4. PMID 19682121
- [Background] Pasina L, Cortesi L, Tiraboschi M, Nobili A, Lanzo G, Tettamanti M, Franchi C, Mannucci PM, Ghidoni S, Assolari A, Brucato A; REPOSI Investigators. Risk factors for three-month mortality after discharge in a cohort of non-oncologic hospitalized elderly patients: Results from the REPOSI study. Arch Gerontol Geriatr. 2018 Jan;74:169-173. doi: 10.1016/j.archger.2017.10.016. PMID 29121542
- [Background] Cao J, Wang T, Li Z, Liu G, Liu Y, Zhu C, Jiao J, Li J, Li F, Liu H, Liu H, Song B, Jin J, Liu Y, Wen X, Cheng S, Wan X, Wu X. Factors associated with death in bedridden patients in China: A longitudinal study. PLoS One. 2020 Jan 29;15(1):e0228423. doi: 10.1371/journal.pone.0228423. eCollection 2020. PMID 31995622
- [Background] Yang SY, Kim ES, Jeon G, Choi KY, Kim JK. Enhanced adhesion of osteoblastic cells on polystyrene films by independent control of surface topography and wettability. Mater Sci Eng C Mater Biol Appl. 2013 Apr 1;33(3):1689-95. doi: 10.1016/j.msec.2012.12.081. Epub 2013 Jan 2. PMID 23827625
- [Background] English KL, Paddon-Jones D. Protecting muscle mass and function in older adults during bed rest. Curr Opin Clin Nutr Metab Care. 2010 Jan;13(1):34-9. doi: 10.1097/MCO.0b013e328333aa66. PMID 19898232
- [Background] Krumholz HM. Post-hospital syndrome--an acquired, transient condition of generalized risk. N Engl J Med. 2013 Jan 10;368(2):100-2. doi: 10.1056/NEJMp1212324. No abstract available. PMID 23301730
- [Background] Drummond MJ, Dickinson JM, Fry CS, Walker DK, Gundermann DM, Reidy PT, Timmerman KL, Markofski MM, Paddon-Jones D, Rasmussen BB, Volpi E. Bed rest impairs skeletal muscle amino acid transporter expression, mTORC1 signaling, and protein synthesis in response to essential amino acids in older adults. Am J Physiol Endocrinol Metab. 2012 May 15;302(9):E1113-22. doi: 10.1152/ajpendo.00603.2011. Epub 2012 Feb 14. PMID 22338078
- [Background] Chizhikov VV, Millen KJ. Control of roof plate development and signaling by Lmx1b in the caudal vertebrate CNS. J Neurosci. 2004 Jun 23;24(25):5694-703. doi: 10.1523/JNEUROSCI.0758-04.2004. PMID 15215291
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] Heit JA, Melton LJ 3rd, Lohse CM, Petterson TM, Silverstein MD, Mohr DN, O'Fallon WM. Incidence of venous thromboembolism in hospitalized patients vs community residents. Mayo Clin Proc. 2001 Nov;76(11):1102-10. doi: 10.4065/76.11.1102. PMID 11702898
- [Background] Heit JA, O'Fallon WM, Petterson TM, Lohse CM, Silverstein MD, Mohr DN, Melton LJ 3rd. Relative impact of risk factors for deep vein thrombosis and pulmonary embolism: a population-based study. Arch Intern Med. 2002 Jun 10;162(11):1245-8. doi: 10.1001/archinte.162.11.1245. PMID 12038942
- [Background] Cohen AT, Tapson VF, Bergmann JF, Goldhaber SZ, Kakkar AK, Deslandes B, Huang W, Zayaruzny M, Emery L, Anderson FA Jr; ENDORSE Investigators. Venous thromboembolism risk and prophylaxis in the acute hospital care setting (ENDORSE study): a multinational cross-sectional study. Lancet. 2008 Feb 2;371(9610):387-94. doi: 10.1016/S0140-6736(08)60202-0. PMID 18242412
- [Background] Zhan C, Miller MR. Excess length of stay, charges, and mortality attributable to medical injuries during hospitalization. JAMA. 2003 Oct 8;290(14):1868-74. doi: 10.1001/jama.290.14.1868. PMID 14532315
- [Background] Hastings SN, Sloane R, Morey MC, Pavon JM, Hoenig H. Assisted early mobility for hospitalized older veterans: preliminary data from the STRIDE program. J Am Geriatr Soc. 2014 Nov;62(11):2180-4. doi: 10.1111/jgs.13095. Epub 2014 Oct 30. PMID 25354909
- [Background] Agmon M, Zisberg A, Gil E, Rand D, Gur-Yaish N, Azriel M. Association Between 900 Steps a Day and Functional Decline in Older Hospitalized Patients. JAMA Intern Med. 2017 Feb 1;177(2):272-274. doi: 10.1001/jamainternmed.2016.7266. No abstract available. PMID 27918776
- [Background] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Background] Binder EF, Schechtman KB, Ehsani AA, Steger-May K, Brown M, Sinacore DR, Yarasheski KE, Holloszy JO. Effects of exercise training on frailty in community-dwelling older adults: results of a randomized, controlled trial. J Am Geriatr Soc. 2002 Dec;50(12):1921-8. doi: 10.1046/j.1532-5415.2002.50601.x. PMID 12473001
- [Background] Daniels R, van Rossum E, de Witte L, Kempen GI, van den Heuvel W. Interventions to prevent disability in frail community-dwelling elderly: a systematic review. BMC Health Serv Res. 2008 Dec 30;8:278. doi: 10.1186/1472-6963-8-278. PMID 19115992